CLINICAL TRIAL: NCT05296200
Title: Cervical Intervertebral Disc Expansion, Vertebral Compliance Reduction and Neck Pain is Induced by 4h of Hyper-buoyancy Flotation That is Only Partially Reversed by 15 Mins 1g Re-loading
Brief Title: Cervical Changes by 4h of Hyper-buoyancy Flotation and Followed by 15 Mins 1g Re-loading
Status: Completed | Type: Observational
Sponsor: Universidad Autonoma de Madrid (Other)
Collaborators: Centro Superior de Estudios Universitarios Lasalle (Unknown)
Responsible Party: Principal Investigator, David Marcos, Principal Investigador, Universidad Autonoma de Madrid
Other Study IDs: CSEULS-PI-032/2020
Record Dates: First submitted 2022-02-23; First posted 2022-03-25 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Intervertebral Disc Herniation; Stiffness; Spine
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observacional group: Subjects must remain to the exposure of gravity (1G) after 4h of hyperbuoyancy floatation(spine unloading)
  Interventions: Device: Hyperbuoyancy Floatation

INTERVENTIONS:
Device: Hyperbuoyancy Floatation — Subjects are laid supine upon a HBF waterbed encased within a wooden frame partially (50%) filled with water (at 36ºC to maintain thermal comfort) super-saturated with magnesium sulphate. Thus, subjects are buoyant, sinking passively into the bed in proportion to their segmental mass.

SUMMARY:
Study with the aim to see the effect on a space ground anaologue, Hyperbuoyancy Floatation (HBF) on cervical column.

DETAILED DESCRIPTION:
the aim of the study is to determine the effect of 4h HBF and subsequent passive 1g axial loading upon stature, cervical IVD height) cervical muscle (Longus Collis and Semispinalis Cervicis) thickness and CSA assessed with ultrasound, cervical vertebral compliance, their relationships to induced stature increments and neck pain.

ELIGIBILITY:
Inclusion Criteria:

* physical requirements (1.57-1.90m, 50-95kg)

Exclusion Criteria:

* current back/neck pain, musculoskeletal disorder, cardiovascular disease, spine surgery and being, or suspected to be pregnant

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: NASA astronaut criteria (1.57-1.90m, 50-95kg)
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2020-03-13 (Actual); Primary Completion 2020-07-25 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Height | up to 2 years
  Standing stature measured by a commercial stadiometer (Seca 217, Germany)

SECONDARY OUTCOMES:
Height of cervical Intervertebral Discs | up to 2 years
  Disc height (C3-T1) measured by ultrasound (Samsung HS40, South Korea)
Longus Collis and Semispinalis Cervicis thickness and cross-sectional area. | up to 2 years
  Neck flexor (Longus Collis) and Neck extensor (Semispinalis Cervicis) were assessed by ultrasound (Samsung HS40, South Korea) and their respective muscle thickness and cross-sectional area was calculated.
Vertebral Stiffness | up to 2 years
  Vertebral stiffness from C0 to L5 was assessed passively (in the prone position) with a handheld differential vertebral compliance transducer (PulStar, Sense Technology Inc., USA) in Newtons.
Self-reported neck pain | up to 2 years
  Pain rating scale (CHAPS) from 0 to 10

CONTACTS AND LOCATIONS:
Overall Officials: Alfonso Gil Martinez, PhD, Study Director — Centro Superior de Estudios Universitarios Lasalle
Locations (1):
- CSEU-Lasalle, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
Data is going to be shared between the investigators authors.

REFERENCES:
- [Background] Green DA, Scott JPR. Spinal Health during Unloading and Reloading Associated with Spaceflight. Front Physiol. 2018 Jan 18;8:1126. doi: 10.3389/fphys.2017.01126. eCollection 2017. PMID 29403389
- [Result] Marshburn TH, Hadfield CA, Sargsyan AE, Garcia K, Ebert D, Dulchavsky SA. New heights in ultrasound: first report of spinal ultrasound from the international space station. J Emerg Med. 2014 Jan;46(1):61-70. doi: 10.1016/j.jemermed.2013.08.001. Epub 2013 Oct 15. PMID 24135505
- [Result] Swanenburg J, Langenfeld A, Easthope CA, Meier ML, Ullrich O, Schweinhardt P. Microgravity and Hypergravity Induced by Parabolic Flight Differently Affect Lumbar Spinal Stiffness. Front Physiol. 2020 Sep 2;11:562557. doi: 10.3389/fphys.2020.562557. eCollection 2020. PMID 32982803
- [Result] McNamara KP, Greene KA, Tooze JA, Dang J, Khattab K, Lenchik L, Weaver AA. Neck Muscle Changes Following Long-Duration Spaceflight. Front Physiol. 2019 Sep 13;10:1115. doi: 10.3389/fphys.2019.01115. eCollection 2019. PMID 31572205